CLINICAL TRIAL: NCT04430075
Title: Transcatheter Repair of Mitral Regurgitation With Edwards PASCAL Transcatheter Valve Repair System: A European Prospective, Multicenter Post Market Clinical Follow-Up (PMCF)
Brief Title: MiCLASP Post Market Clinical Follow-Up (PMCF) Study
Acronym: MiCLASP
Status: Recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-08
Record Dates: First submitted 2019-12-19; First posted 2020-06-12 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Mitral Regurgitation; Mitral Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Edwards PASCAL Transcatheter Valve Repair System and Edwards PASCAL Precision Transcatheter Valve Repair System — Transcatheter Valve Repair with Edwards PASCAL and PASCAL Precision System

SUMMARY:
This is a postmarket clinical follow up study on the safety and effectiveness of the Edwards PASCAL Transcatheter Valve Repair System and the Edwards PASCAL Precision Transcatheter Valve Repair System in transcatheter mitral valve repair.

DETAILED DESCRIPTION:
The objectives of this clinical study are to collect data on the safety of the Edwards PASCAL Transcatheter Valve Repair System and the Edwards PASCAL Precision Transcatheter Valve Repair System in transcatheter mitral valve repair and on the effectiveness of the Edwards PASCAL System and Edwards PASCAL Precision System in improving MR, functional status and quality of life in a post market setting.

ELIGIBILITY:
Inclusion Criteria:

1. Mitral TEER patients eligible per the current approved indication after Heart Team discussion and agreement
2. Patient is willing and able to attend all follow-up visits and to perform all tests
3. Provision of written informed consent

Exclusion Criteria:

1. Patients are not eligible per the current Instructions for Use
2. Non-elective or emergency TEER procedure for mitral regurgitation
3. Patients in ICU prior to the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at or over the age of 18 determined to require percutaneous reconstruction of an insufficient mitral valve [MR ≥ 2+ (PASCAL patients) or MR ≥ 3+ (PASCAL Precision patients)] by a Heart Team who assesses patient risk and anatomic suitability should be considered for inclusion in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with major adverse events (MAE rates) | 30 days
  The primary safety endpoint is the proportion of patients with major adverse events (MAEs) at 30 days
Change in mitral regurgitation severity (scale of 0-4+) by echocardiography | Discharge: defined as discharge or 7 days post-procedure, whichever comes first
  Mitral regurgitation severity will be assessed by echocardiography at timepoint discharge on a scale from 0-4+ and compared to timepoint baseline Mitral regurgitation severity

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Lurz, Prof.Dr.med., Principal Investigator — Johannes Gutenberg University Mainz
Locations (36):
- Medizinische Universität Wien/AKH Wien, Vienna, Austria
- Germany (25):
  - Universitäts-Herzzentrum Freiburg Campus Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Universität Tuebingen, Tübingen, Baden-Wurttemberg
  - Uniklinikum Ulm, Ulm, Baden-Wurttemberg
  - Uniklinikum Erlangen, Erlangen, Bavaria
  - Medizinische Klinik I- Campus Grosshadern, München, Bavaria
  - Immanuel Klinikum Bernau, Bernau bei Berlin, Brandenburg
  - Universitätsklinikum Giessen UKGM, Giessen, Hesse
  - Universitaeres Herzzentrum Goettingen, Göttingen, Lower Saxony
  - Westdeutsches Herzzentrum / Uniklinik Essen, Essen, Nordrhine Westfalia
  - Contilia Herz- und Gefäßzentrum,Elisabeth-Krankenhaus Essen, Essen, Nordrhine Westfalia
  - Herz- und Diabeteszentrum NRW - Bad Oeynhausen, Bad Oeynhausen, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Herzzentrum Universitaetsklinik Herzzentrum Universitaetsklinik Cologne, Cologne, North Rhine-Westphalia
  - St.-Johannes-Hospital, Dortmund, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, North Rhine-Westphalia
  - Helios Klinikum Siegburg, Siegburg, North Rhine-Westphalia
  - Herzzentrum Universitätsklinik Dresden, Dresden, Saxony
  - Universitäres Herzzentrum Lübeck, Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Charité Berlin, Berlin
  - MVZ-CCB, Frankfurt
  - Universitares Herzzentrum Hamburg, Hamburg
  - Kath. Marienkrankenhaus Hamburg GmbH, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Heart Centre of the University Leipzig, Leipzig
- Hygeia Hospital, Athens, Greece
- Italy (3):
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Ospedale del Cuore G. Pasquinucci Massa, Massa
  - IRCCS Policlinico San Donato, San Donato Milanese
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC, Rotterdam
- The Cardinal Stefan Wyszyński, Institute of Cardiology, Warsaw, Poland
- Hospital Alvaro Cunqueiro, Vigo, Spain
- Inselspital Bern, Bern, Switzerland
- Wythenshawe Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No